CLINICAL TRIAL: NCT06506409
Title: Effectiveness of Smart-Video Based Game Therapy and Otago-Based Structured Exercises in Women With Osteoporosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Yağmur KARAMAN POLAT, Research Assistant, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedipolU-FTR-YKP-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Osteoporosis
Keywords: game therapy; rehabilitative game; otago exercise
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: We have three parallel groups: Two treatment groups and one control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Smart-Video Based Game Therapy Group (Active Comparator): The Active Arcade program will be practiced 2 days a week for 8 weeks. Individuals in this group will be given a 1-minute rest break between games. Sessions will be approximately 30 minutes. The selected games focus on balance, coordination and weight transfer.
  Interventions: Device: Smart-Video Based Game Therapy
- Otago Based Structured Exercise Group (Active Comparator): Exercises will be done 2 days a week for 8 weeks and last approximately 30 minutes. In general, if individuals can perform 2 sets of 10 repetitions of movements at a difficulty level with quality, they can move on to a higher difficulty level. It consists of warm-up, balance and strengthening exercises. It was developed to increase balance.
  Interventions: Other: Otago Based Structured Exercise
- Control group (Active Comparator): A training presentation based on the guidelines and individuals' needs will be developed for participants in the control group. The presentation will include an infographic developed with the CANVA program, a test created with Google Forms, and a summary video developed with the Powtoon program. The created presentation will be presented online to individuals in the control group, and the participants will be followed by phone once a week for 8 weeks. The topics of the training will be: What is Osteoporosis, Osteoporosis Prevalence, Findings and Risk Factors, Diagnosis of Osteoporosis, Osteoporosis Prevention and Nutrition, Osteoporosis and Exercise, Preventing Falls.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Smart-Video Based Game Therapy — The Active Arcade program will be practiced 2 days a week for 8 weeks. Individuals in this group will be given a 1-minute rest break between games. Sessions will be approximately 30 minutes. Selected games focus on balance, coordination and weight transfer.
  Arms: Group 1: Smart-Video Based Game Therapy Group
Other: Otago Based Structured Exercise — Exercises will be done 2 days a week for 8 weeks and last approximately 30 minutes. In general, if individuals can perform 2 sets of 10 repetitions at a difficulty level with quality, they can move on to a higher difficulty level. It consists of warm-up, balance and strengthening exercises. It was developed to increase balance.
  Arms: Otago Based Structured Exercise Group
Other: No intervention — A training presentation based on the guidelines and individuals' needs will be developed for participants in the control group. The presentation will include an infographic developed with the CANVA program, a test created with Google Forms, and a summary video developed with the Powtoon program. The created presentation will be presented online to individuals in the control group, and the participants will be followed by phone once a week for 8 weeks. The topics of the training will be: What is Osteoporosis, Osteoporosis Prevalence, Findings and Risk Factors, Diagnosis of Osteoporosis, Osteoporosis Prevention and Nutrition, Osteoporosis and Exercise, Preventing Falls.
  Arms: Control group

SUMMARY:
In this project, researchers evaluated the effects and differences of smart-video based game therapy and Otago-based structured exercises in women with osteoporosis; aimed to evaluate their applicability in women with osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a musculoskeletal disease characterized by decreased bone mass and deterioration of the microstructure of the bone. The aim of the study is to use smart-based video-based play therapy and Otago-based structured exercises in women with osteoporosis; To evaluate the effect on bone quality, lower extremity muscle strength, balance, fear of falling, kinesiophobia and quality of life.

Working Groups Group 1: Smart Based Video Based Game Therapy Group Group 2: Otago Based Structured Exercise Group Group 3: Control Group Participants who agree to participate in the study are first evaluated with the Mental State Assessment - Standardized Mini Mental Test and Game Therapy group with the Simulator Illness Questionnaire and System Usability Scale, and if they meet the participation criteria, our study involves face-to-face interviews and blood and urine samples are routinely performed by the doctor on all patients at their first visit. Bone quality will be evaluated using bone turnover markers. Static balance with Romberg Test, dynamic balance with Four Square Step Test, functionality with Timed Up and Go Test, fear of falling with International Fall Activity Scale, kinesiophobia with Tampa Kinesiophobia Scale, muscle strength with Myometer, quality life with European Osteoporosis Association Quality of Life Questionnaire-41 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women in the climacteric period with osteoporosis between the ages of 45-65
* Those with DEXA T score < -2.5 SD,
* Those who have independent ambulation,
* Those who have no history of falling in the last year
* Those with a mini mental test score of 24 and above

Exclusion Criteria:

* Those who have participated in any exercise program in the last 3 months,
* Those who need support in ambulation,
* Those with a history of pathological fracture due to significant post-traumatic or malignancy,
* Those who have any systemic disease that may hinder the practices,
* Those with vestibular dysfunction,
* For participants in the smart video-based game therapy group, those who are not suitable to use the system according to the System Usability Scale and Simulator Illness Questionnaire

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in the climacteric period with osteoporosis
Enrollment: 51 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
blood and urine samples | eight weeks
  Evaluation will be made with Bone turnover markers in the individuals' blood and urine samples. Bone turnover markers are classified as bone formation and resorption markers. Bone formation markers; serum osteocalcin (OC), serum total alkaline phosphatase (ALP); Bone resorption markers; urine deoxypyridinoline (DPD), free collagen cross-linked N-telopeptide (NTX).
Romberg test | eight weeks
  It will be evaluated with the Romberg test. It is desirable to maintain postural control for 20-30 seconds with feet together, eyes open and closed. Additionally, the Romberg test is performed on a soft ground.
Four Square Step Test | eight weeks
  It will be evaluated with the Four Square Step Test. By placing two canes on a flat surface, 4 squares are created and the squares are numbered. The participant is told that he/she must step into each square in the successive order (1-2-3-4-1-4-3-2-1) as fast as possible, without touching the canes, and that both feet must contact the ground in each square. The time to complete the sequence is recorded as a score. 2 scores are measured and the best one is taken.
time up and go test | eight weeks
  Evaluation will be made with a time up and go test. A point is marked 3 m away from the chair where the participant is sitting. The participant is asked to get up from the chair, walk 3 m, turn back and sit on the chair again, and the time to complete the test is measured and recorded in seconds.
International Falls Effectiveness Scale | eight weeks
  It will be evaluated with the International Falls Effectiveness Scale. It is a scale that evaluates how confident elderly individuals are in their daily life activities and shows their level of fear of falling. Each item of the scale, which consists of 16 items, is rated between 1 and 4 points (I am not worried at all: 1 point, I am a little worried: 2 points, I am quite worried: 3 points, I am very worried: 4 points). The total scale score ranges from 16 to 64, with a higher score indicating increased fear of falling.
Tampa Kinesiophobia Scale | eight weeks
  The Tampa Kinesiophobia Scale developed by Miller, Kori and Todd will be used to evaluate kinesiophobia. It consists of 17 items including parameters of injury, re-injury, fear and avoidance in work-related activities. The scale uses a 4-point system, where 1 point means strongly disagree and 4 points means completely agree. A high score from the scale indicates a high kinesiophobia valu
myometer | eight weeks
  The lower extremity muscle strength of all participants will be measured with a myometer. Muscle groups to be evaluated: Gluteus medius, gluteus maximus, adductor, quadriceps femoris, hamstring, gastrocnemius-soleus, tibialis anterior. Each measurement is repeated 3 times and the average of the test is recorded in kilograms.
European Osteoporosis Association Quality of Life Questionnaire-41 | eight weeks
  European Osteoporosis Association Quality of Life Questionnaire-41, such as pain (5 items), physical function (17 items), social activity (7 items), general health assessment (3 items) and mental function (9 items); It consists of 5 subscales examining five dimensions of health. It is scored on a 1-5 Likert type scale. A high score indicates poor quality of life.

SECONDARY OUTCOMES:
Standardized Mini Mental Test | eight weeks
  Standardized Mini Mental Test (MMSE) will be used to evaluate mental status. MMSE can be used to screen for cognitive impairment, estimate the severity of cognitive impairment at a particular point in time, track the course of cognitive changes in the individual over time, and evaluate the individual's response. It evaluates different cognitive status subheadings such as attention, language, memory, orientation, and visual spatial competence. MMSE is scored between 0-30 and >24 is interpreted as normal cognitive status.
Simulator Sickness Survey | eight weeks
  Simulator Sickness Survey; 16 symptoms, such as eye fatigue, nausea, sweating and headache, are evaluated in 4 different severity levels (none, mild, moderate and severe). Symptoms; They are grouped into three categories: nausea, oculomotor disturbance and disorientation. Higher scores in each category indicate stronger disease symptoms.
System Usability Scale | eight weeks
  It consists of 10 statements that help evaluate the ease of use of websites, software, hardware, mobile devices and other technological applications. The scale, which uses a 5-point Likert scale, is basically a survey created to evaluate usability. The average value is taken as 68, and a score greater than 68 indicates that the system is above average. Products with the highest usability evaluation are in the A+ class and the percentage range is between 96-100.

CONTACTS AND LOCATIONS:
Locations (1):
- Ümraniye Eğitim Araştırma Hastanesi, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No